CLINICAL TRIAL: NCT02141009
Title: Response to Pneumococcal Vaccination in Patients After Community Acquired Pneumonia With Streptococcus Pneumoniae Compared to Pneumonia Patients With Another Pathogen.
Brief Title: Community Acquired Pneumonia: Outcome, Quality of Life and Immune Status
Acronym: CAPolista
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Gertjan Wagenvoort, MD, St. Antonius Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL44924.100.13; 2013-002166-39 (EudraCT Number)
Record Dates: First submitted 2014-05-13; First posted 2014-05-16 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Pneumonia; Streptococcus Pneumoniae; Immune Response
Keywords: Vaccination, prevnar, PCV13
MeSH Terms: conditions — Pneumonia | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prevnar 13 (Other): Prevnar 13, 1 administration of 1 single dose (0.5mL)
  Interventions: Biological: Prevnar 13

INTERVENTIONS:
Biological: Prevnar 13
  Other Names: Prevenar 13; pneumococcal 13-valent conjugate vaccin; PCV13

SUMMARY:
Community acquired pneumonia (CAP) is an important health problem with significant morbidity, mortality and cost. The most identified pathogen in CAP is Streptococcus pneumoniae. This was also the causative agent most frequently found in the Ovidius and Triple-P study, two consecutive clinical trials initiated by the St. Antonius Hospital Nieuwegein. Diagnosis of pneumococcal pneumonia can be based on positive blood cultures, sputum cultures, urine antigen testing or a serotype specific antibody response. When pneumococcal pneumonia is diagnosed by a positive culture, a matching serotype specific antibody response is expected. However not all patients in the Ovidius and Triple-P study with a culture proven pneumococcal pneumonia showed an antibody response against the infecting pneumococcal serotype. Patients who survived pneumococcal pneumonia are considered as a high-risk population for pneumococcal disease in the future. Possibly these patients have an impaired immune response against S. pneumoniae. In this study, pneumococcal vaccination of patients with S. pneumoniae CAP in the past enables investigating their immune response after vaccination compared to patients with CAP due another causative agent. Furthermore this study provides information to determine if there is a difference in vaccination response between pneumococcal pneumonia patients who had a culture matching serotype specific antibody response and between pneumococcal pneumonia patients who failed to elicit this response previously. Possibly these latter patients had a temporarily low titre due to the infection but another explanation is that there might be a structurally impaired immune response against S. pneumoniae or certain serotypes.

DETAILED DESCRIPTION:
1. Introduction & rationale Community acquired pneumonia (CAP) is an important health problem with significant morbidity, mortality and cost. It is one of the main causes of disease and death worldwide and causes the most deaths by infection in the United States. Streptococcus pneumoniae is the most commonly identified pathogen in CAP.(1)

   S. pneumoniae is a gram-positive, alpha haemolytic bacterium that is surrounded by an external polysaccharide capsule. There is a difference in composition of this capsule between the 92 different serotypes of S. pneumoniae. Each serotype differs in virulence and prevalence. The external polysaccharide capsule is the main trigger for the specific antibody response and is the basis for pneumococcal vaccines. As it is impossible to develop a vaccine that protects children, immune compromised adults and older adults to all serotypes, the vaccines are based on the most common and virulent serotypes.

   Nowadays a 13-valent pneumococcal conjugate vaccine, Prevnar 13 (PCV13), is used widely to vaccinate children. This vaccine contains the seven serotypes present in PCV7 (4, 6B, 9V, 14, 18C, 19F and 23F) plus the emerging serotypes 1, 3, 5, 6A, 7F and 19A.(2) In the Netherlands however the 10-valent pneumococcal conjugate vaccine, Synflorix (PCV10), is still used to vaccinate children in the national infant vaccination.(3)

   Van Mens et al investigated the contribution of S. pneumoniae in CAP by measuring serologic responses in patients who were hospitalized due to CAP in the Ovidius and Triple P study, two consecutive clinical trials initiated by the St Antonius Hospital Nieuwegein. This analysis showed a much higher proportion of patients with pneumococcal pneumonia than was diagnosed by conventional methods alone (i.e. blood cultures, sputum cultures or urine antigen tests). Interestingly some patients with a culture proven pneumococcal pneumonia did not show a serotype specific antibody response to the infecting serotype.(4) Possibly these patients had a temporarily low titre due to the infection but another explanation is that there might be a structurally impaired immune response against S. pneumoniae or certain serotypes.

   Borrow et al vaccinated 107 children with PCV7 after invasive pneumococcal disease (IPD) following a routine infant immunization schedule. Pneumococcal serotype specific antibody measurements were performed and showed failure to respond to the infecting serotype in 8 children, even though these children received 2 or more doses of PCV. Two children failed to respond to a serotype different than the infecting serotype.(5)

   In this study the humoral and cellular immune response after vaccination with Prevnar 13 will be measured in patients who have had CAP with S. pneumoniae. The patients will be recruited from the Ovidius and Triple-P study, two consecutive clinical trials initiated by the St. Antonius Hospital Nieuwegein.(6,7) Patients who survived pneumococcal pneumonia are considered as a high-risk population for pneumococcal disease in the future.(8) Possibly these patients have less response to pneumococcal vaccination because of an impaired immune response against S. pneumoniae. Special interest goes to vaccination responses in the subgroup of pneumococcal pneumonia patients without a culture matching specific antibody response in order to investigate if this reflects the failure to elicit an immune response during pneumonia found by Van Mens et al.
2. Objectives

   Primary Objective:

   • To investigate antibody response after pneumococcal vaccination in patients with community acquired pneumococcal pneumonia compared to pneumonia patients with another pathogen.

   Secondary Objective(s):
   * To investigate antibody response after pneumococcal vaccination in patients with community acquired pneumococcal pneumonia who failed to elicit a specific antibody response.
   * To investigate the cellular immune responses after pneumococcal vaccination in patients with community acquired pneumococcal pneumonia in the past compared to pneumonia patients with another pathogen.
   * To investigate quality of life by the RAND-36 score in patients with community acquired pneumococcal pneumonia compared to pneumonia patients with another pathogen.
   * To investigate the long-term mortality after community acquired pneumococcal pneumonia.
3. Study design The design is a prospective cohort study in which response to pneumococcal vaccination and immune function after CAP with S. pneumoniae will be investigated. Patients who were included in the Ovidius or Triple-P study and diagnosed with pneumococcal pneumonia (with cultures, urine antigen test or serology) will be included. The control group will consist of patients who were included in the Ovidius or Triple-P study and diagnosed with community acquired pneumonia with another pathogen.
4. Working plan All patients and controls will receive vaccination with Prevnar 13. During this visit information about the medical history, medication usage and daily status will be obtained. Patients are also asked to fill-in a quality of life questionnaire (RAND-36; section F Questionnaires). Sera will be obtained before vaccination and three - four weeks after vaccination to determine antibody response against different serotypes of S. pneumoniae. The study will end with the last visit of the last patient; the duration of the study will be approximately 2 months (dependent on the moment of inclusion of the patient).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who participated in the Ovidius or Triple-P study (2004-2009).
2. Diagnosis in these studies with pneumococcal pneumonia or pneumonia due another identified organism.
3. Age ≥ 18 years.
4. Signing of informed consent.

Exclusion Criteria:

1. Diagnosis of pneumonia without an identified causative organism.
2. Fever at time of vaccination.
3. Previous/known allergic reaction to any of the components of the vaccine given.
4. Mentally incompetent.
5. Previous pneumococcal conjugate vaccination.
6. Pneumococcal polysaccharide vaccination within 6 months prior to inclusion.
7. Clinical pneumonia within 1 month prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Antibody titers against pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F | Change in antibody titers week 1 and week 3-4
  Antibody titers against pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F and avidity maturation will be determined using Luminex technology.
  A serotype specific response to vaccination is defined as a ≥ 2-4-fold increase in serum antibody titre from baseline (and a post vaccination titer > 0.35 µg/mL) or a post immunization titer ≥ 1.3 ug/mL

SECONDARY OUTCOMES:
Antibody avidity maturation against pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F | Change in avidity between week 1 and week 3-4
  Antibody avidity maturation against pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F will be determined using Luminex technology in combination with a chaotropic agent.
  The avidity maturation will be calculated with relative avidity index (RAI) in percent based on baseline and post vaccination measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Ger T Rijkers, Prof, Study Director — St. Antonius Hospital; Gertjan H Wagenvoort, MD, Principal Investigator — St. Antonius Hospital; Bart JM Vlaminckx, Phd, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Hospital Nieuwegein, Nieuwegein, Utrecht, Netherlands

REFERENCES:
- [Background] File TM. Community-acquired pneumonia. Lancet. 2003 Dec 13;362(9400):1991-2001. doi: 10.1016/S0140-6736(03)15021-0. PMID 14683661
- [Background] Principi N, Esposito S. Use of the 13-valent pneumococcal conjugate vaccine in infants and young children. Expert Opin Biol Ther. 2012 May;12(5):641-8. doi: 10.1517/14712598.2012.670217. Epub 2012 Mar 7. PMID 22397739
- [Background] van Mens SP, Meijvis SC, Endeman H, van Velzen-Blad H, Biesma DH, Grutters JC, Vlaminckx BJ, Rijkers GT. Longitudinal analysis of pneumococcal antibodies during community-acquired pneumonia reveals a much higher involvement of Streptococcus pneumoniae than estimated by conventional methods alone. Clin Vaccine Immunol. 2011 May;18(5):796-801. doi: 10.1128/CVI.00007-11. Epub 2011 Mar 2. PMID 21367978
- [Background] Borrow R, Stanford E, Waight P, Helbert M, Balmer P, Warrington R, Slack M, George R, Miller E. Serotype-specific immune unresponsiveness to pneumococcal conjugate vaccine following invasive pneumococcal disease. Infect Immun. 2008 Nov;76(11):5305-9. doi: 10.1128/IAI.00796-08. Epub 2008 Sep 8. PMID 18779338
- [Background] Endeman H, Meijvis SC, Rijkers GT, van Velzen-Blad H, van Moorsel CH, Grutters JC, Biesma DH. Systemic cytokine response in patients with community-acquired pneumonia. Eur Respir J. 2011 Jun;37(6):1431-8. doi: 10.1183/09031936.00074410. Epub 2010 Sep 30. PMID 20884746
- [Background] Meijvis SC, Hardeman H, Remmelts HH, Heijligenberg R, Rijkers GT, van Velzen-Blad H, Voorn GP, van de Garde EM, Endeman H, Grutters JC, Bos WJ, Biesma DH. Dexamethasone and length of hospital stay in patients with community-acquired pneumonia: a randomised, double-blind, placebo-controlled trial. Lancet. 2011 Jun 11;377(9782):2023-30. doi: 10.1016/S0140-6736(11)60607-7. Epub 2011 Jun 1. PMID 21636122
- [Background] Restrepo MI, Faverio P, Anzueto A. Long-term prognosis in community-acquired pneumonia. Curr Opin Infect Dis. 2013 Apr;26(2):151-8. doi: 10.1097/QCO.0b013e32835ebc6d. PMID 23426328
- [Background] Paris K, Sorensen RU. Assessment and clinical interpretation of polysaccharide antibody responses. Ann Allergy Asthma Immunol. 2007 Nov;99(5):462-4. doi: 10.1016/S1081-1206(10)60572-8. PMID 18051217
- [Derived] Wagenvoort GHJ, Vlaminckx BJM, van Kessel DA, Geever RCL, de Jong BAW, Grutters JC, Bos WJW, Meek B, Rijkers GT. Pneumococcal conjugate vaccination response in patients after community-acquired pneumonia, differences in patients with S. pneumoniae versus other pathogens. Vaccine. 2017 Sep 5;35(37):4886-4895. doi: 10.1016/j.vaccine.2017.07.088. Epub 2017 Aug 9. PMID 28802755